CLINICAL TRIAL: NCT00895648
Title: Phase II Study of Neo-adjuvant Pemetrexed (ALIMTA) Plus Cisplatin Followed by Surgery and Radiation Therapy for Malignant Pleural Mesothelioma
Brief Title: Pemetrexed (ALIMTA) Plus Cisplatin Followed by Surgery and Radiation Therapy for Mesothelioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual due to competing study for same group of patients
Sponsor: University Health Network, Toronto (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-0815-C
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Mesothelioma; Pleural Mesothelioma
Keywords: Meso; mesothelioma; pleura; pleural
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alimta plus Cisplatin (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m² iv infusion every 3 weeks for 3 cycles
  Other Names: Alimta
Drug: Cisplatin — 75 mg/m² iv infusion every 3 weeks for 3 cycles

SUMMARY:
Despite the best surgical efforts, complete removal of mesothelioma is possible in approximately 30% of the patients. When surgical removal is complete, chemotherapy followed by radiation therapy is recommended as an effort to improve control over the cancer and survival. This combination of treatments is called TRIMODALITY therapy. Unfortunately, the chances for the tumor coming back after TRIMODALITY therapy remains high. When surgical removal is not complete or not possible, some patients may receive chemo and/or radiation therapy to achieve control over the cancer, but the chances of tumor to growth again remains high and the chances of long term survival remains low.

The combination of Pemetrexed (Alimta) with Cisplatin has been approved as one of the standard chemotherapy drug combinations for the treatment in advanced Malignant Pleural Mesothelioma, and there is likely a group of patients who may benefit and potentially be cured by this therapy. In an effort to achieve a better chance of complete removal of the cancer and long term survival, the investigators are interested in using this drug combination of Pemetrexed + Cisplatin before surgery and offer radiation therapy after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of MPM stages I to III. Patients will be clinically staged using the AJCC/UICC TNM staging criteria (see Protocol Appendix 2). Eligible stages:

   * Patients must be M0.
   * Patients with T1, T2, and T3 disease (without cardiac involvement) are eligible. T status can be established clinically and radiologically or at exploratory thoracotomy without surgical resection.
   * Patients with N0, N1, or N2 disease are eligible.
2. Performance status of 0 to 2 on the ECOG performance status schedule. See protocol Appendix 3
3. No prior systemic chemotherapy. No prior intracavitary cytotoxic drugs or immunomodulators, unless given for the purpose of chemical pleurodesis.
4. No previous surgical procedure for mesothelioma, with the exception of previous chemical pleurodesis and biopsy.
5. No previous radiation therapy for mesothelioma, or to the thorax.
6. Patients must be judged to be suitable candidates for this therapy at the UHN by the attending medical oncologist, thoracic surgeon, and radiation oncologist before enrolment.
7. Estimated life expectancy of at least 12 weeks.
8. Adequate organ function including the following:

   * Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) ³1,500/uL , platelets ³100,000/uL, hemoglobin ³ 9g/dL
   * Hepatic: bilirubin £1.5 times institutional upper limit of normal, alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) £3 times institutional upper limit of normal
   * Renal: Creatinine £1.5 times institutional upper limit of normal; or Creatinine clearance ³50 mL/min/1.73 m² for patients with creatinine levels above institutional normal upper limit level. Cockcrot and Gault formula Appendix 4.
   * Pulmonary function tests:

   Predicted post-operative DLCO (ppoDLCO) of > 35%.

   If the ppoDLCO is </= 35%, then additional studies will be done to determine the patient's ability to tolerate the resection. The surgeon will correlate these results with the patient's clinical status and make a decision as to the feasibility of resection.
9. Female patients of childbearing potential must test negative for pregnancy at the time of enrolment based on a serum pregnancy test. Male and female patients must agree to use a reliable method of birth control during and for 3 months following the last dose of radiation therapy.
10. Patients must sign an informed consent

Exclusion Criteria:

1. Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
2. Have previously completed or withdrawn from this study or any other study investigating pemetrexed
3. Pregnancy or breast-feeding.
4. Serious concomitant systemic disorders (e.g., active infection) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
5. Second active primary malignancy except in situ carcinoma of the cervix, adequately treated non-melanomatous carcinoma of the skin, low grade (Gleason score < 6) localized adenocarcinoma of the prostate or other malignancy treated at least 2 years previously with no evidence of recurrence.
6. Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents for a 5-day period (8 day period for long-acting agents such as piroxicam).
7. Inability or unwillingness to take folic acid, vitamin B12 supplementation, or dexamethasone.
8. Refusal to have any of the treatment in the protocol (chemotherapy, extrapleural pneumonectomy, and radiation therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
median relapse-free survival (RFS) | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Ron Feld, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada